CLINICAL TRIAL: NCT01729975
Title: Comparative Study of Specular Microscopes for the Measurement of Endothelial Cell Densities, Coefficient of Variation of Endothelial Cell Area, ％Hexagonality, and Central Corneal Thickness
Brief Title: Comparative Study of Specular Microscope for Cell Density, Coefficient of Variation, Hexagonality and Corneal Thickness
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: CEM-530-US-001
Record Dates: First submitted 2012-11-07; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Corneal and Endothelial Cell Measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 18-28 years old Non-pathologic
- 29-80 years old Non-Pathologic
- 29-80 years old pathologic corneal disease

SUMMARY:
The primary objective of this clinical study is to collect clinical data to support an FDA 510(k) submission for the Nidek Specular Microscope CEM-530. The secondary objective is to evaluate any adverse events found during the clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Non-Pathologic: Male or female subjects from 18 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed. Subjects who follow the instructions by Principal/Clinical investigator or clinical staff at the clinical site, and can visit on a scheduled examination date.
* Pathologic: Male and female subjects from 29 to 80 years old who have full legal capacity to volunteer on the date the informed consent is signed. Subjects who follow the instructions by Principal/Clinical investigator or clinical staff at the clinical site, and can visit on a scheduled examination date and subjects who have any of the following conditions:

  * History of Post-op surgical trauma including, Psudophakic or Aphakic blous keratopathy or glaucoma surgery
  * History of corneal transplant
  * Physical injury or trauma to the cornea
  * Long term Fuch's dystrophy/Guttata (and other corneal endothelial dystrophy)
  * Keratoconus
  * Long term PMMA contact lens use

Exclusion Criteria:

* Non-Pathologic subjects who have the following conditions:

  * Long term Diabetes
  * Dementia
  * Subjects who have other life threatening and/or debilitating systemic diseases
  * History of corneal transplant
  * Long term Fuch's dystrophy (and other corneal endothelial dystrophy)
  * Keratoconus
  * Guttata
  * Diabetic retinopathy
  * History of cataract or ocular surgical procedures that render the cornea opaque or otherwise impact its ability to be imaged using the investigational device.
  * All contact lens wearers
* Pathologic subjects who have Dementia or who have other life threatening and/or debilitating systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology Practice
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Corneal and Endothelial Cell Measurements | single time point - 1 day
  Substantial equivalence to a predicate device with respect to corneal and endothelial cell measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States